CLINICAL TRIAL: NCT04640974
Title: A Prospective Study of a Single Injection Cross-linked Sodium Hyaluronate Combined With Triamcinolone Hexacetonide (CINGAL®) to Provide Symptomatic Relief of Osteoarthritis of Ankle Joint
Brief Title: Study of Cingal® for Symptomatic Relief of Osteoarthritis of Ankle Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cingal 20-03
Record Dates: First submitted 2020-11-19; First posted 2020-11-23 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis, Ankle
Keywords: Sodium Hyaluronate; Triamcinolone Hexacetonide
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cingal (Experimental): Single injection of Cingal into the ankle joint of subjects diagnosed with osteoarthritis of the ankle.
  Interventions: Device: Cingal

INTERVENTIONS:
Device: Cingal — Single injection into the ankle joint of a 4 ml unit dose of Cingal containing 88 mg (22 mg/ml) of cross-linked sodium hyaluronate and 18 mg (4.5 mg/ml) of triamcinolone hexacetonide (TH).

SUMMARY:
This Trial will obtain clinical data to support an expanded indication for a single injection of Cingal® used for the symptomatic relief of osteoarthritis in the ankle joint.

DETAILED DESCRIPTION:
Single injection into the ankle joint of a 4 ml unit dose of Cingal containing 88 mg (22 mg/ml) of cross-linked sodium hyaluronate and 18 mg (4.5 mg/ml) of triamcinolone hexacetonide (TH).

ELIGIBILITY:
Screening Inclusion Criteria:

1. Age 18 years or older
2. Body Mass Index (BMI) ≤ 35 kg/m2
3. Diagnosis of symptomatic osteoarthritic joint in the index ankle (Kellgren-Lawrence grade I to III) to be treated with Cingal injection.
4. Failed conservative treatment for joint osteoarthritis.
5. NRS pain on walking ≥4 and ≤9 in the index ankle.
6. Subject must be willing to abstain from other treatments of the index ankle for the duration of the study.
7. Subject is willing to discontinue all analgesics including NSAIDs, except acetaminophen/paracetamol, at least seven days before the treatment injection and through the completion of the study.
8. Subject is willing to use only acetaminophen/paracetamol (up to a maximum of 4.0 grams per day per the package insert) for the treatment of joint pain for the duration of the study. At least forty-eight hours prior to the Baseline Visit and each follow-up visit, the subject is willing to discontinue use of acetaminophen/paracetamol.
9. Subject is willing to maintain a stable dose of oral glucosamine and/or chondroitin sulfate products throughout the study, if taken prior to signing the informed consent form (ICF).
10. Able and willing to provide signed informed consent

Baseline Inclusion Criteria

1. NRS pain on walking ≥4 and ≤ 9 in index ankle

Screening Exclusion Criteria:

1. History of hypersensitivity to any of the ingredients in the hyaluronan or corticosteroids
2. Infection or skin disease in the area of the injection site or ankle joint
3. NRS pain on walking > 3 in the contralateral ankle
4. NRS pain on walking > 3 in the ipsilateral knee or hip
5. Subject received an injection of Hyaluronic Acid (HA) and/or steroid in either ankle within 6 months of signing the informed consent form (ICF). A subject will be excluded if they are planning to receive an HA or steroid injection (other than the study injection) in either ankle during the course of this study.
6. Known inflammatory or autoimmune disorders (including rheumatoid arthritis, gout), or other pre-existing medical conditions that, in the opinion of the investigator, could impact treatment of the index ankle or affect the ability of the subject to accurately complete the study questionnaires and comply with the study requirements.
7. Subject is taking medications at the time of signing the ICF which could interfere with the treatment procedure, healing and/or assessments. This includes but is not limited to oral or injectable anticoagulant treatments, anti-aggregant platelet treatment, chronic opioid analgesics. Low dose aspirin used for cardiovascular protection is allowed if a stable regimen is maintained for the duration of the study.
8. Subjects who had an oral, intramuscular, intravenous, rectal suppository or topical (excluded in index ankle only) corticosteroid prior 30 days of signing the ICF are excluded. Topical corticosteroid use at any site other than the index ankle is allowed.
9. Significant trauma to the index ankle within 26 weeks of screening
10. Chronic use of narcotics or cannabis.
11. Ligament instability or tear in index ankle.
12. Chronic impingement in the index ankle requiring surgical treatment
13. Diagnosis of fibromyalgia
14. Diagnosis of osteonecrosis in index ankle
15. Subject has significant varus or valgus deformity greater than 10 degrees in either knee.
16. Subject requires consistent use of an assistive device (e.g. wheelchair, walker, etc.) Occasional use of a cane is acceptable.
17. Uncontrolled diabetes with HbA1c of >7%.
18. Subject is a woman who is pregnant or breastfeeding at the Screening Visit or a woman of child bearing potential who refuses to use effective contraception during the course of the study.
19. Subject is receiving or in litigation for worker's compensation.
20. Otherwise determined by the investigator to be medically unsuitable for participation in this study.

Baseline Exclusion Criteria

1. Subject has a decrease of ≥ 2 in the NRS pain on walking from Screening to Baseline in the index ankle.
2. Subject has a contraindication to continue with the study treatment injection based on the visual appearance of the synovial fluid aspirate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara Mezger, Study Director — Anika Therapeutics
Locations (4):
- Krajská zdravotní, a.s. - Masarykova nemocnice Ústí nad Labem, o.z., Ústí nad Labem, Czechia
- Poland (3):
  - NZOZ MEDI-SPATZ M.Spatz, Gliwice
  - SPORTO sp. z o.o, Lodz
  - Przychodnia Rodzinna na Sadowej, Torun

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cingal
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cingal
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.12 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 1
  Unknown or Not Reported | 0
Index Ankle [Count of Participants; unit: Participants]
  Right | 16
  Left | 9

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (NRS) Pain on Walking
Description: Reduction of Index Ankle Numerical Rating Scale (NRS) Pain on Walking from baseline to 6 months post injection was obtained from participant responses. The NRS Pain Score ranged from 0 = No Pain to 10 = Worst Pain Level. A negative value for the change in Pain Score indicates less pain post-treatment. A larger negative value indicates a higher level of improvement, and a better outcome.
Time Frame: 6 months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cingal
Number analyzed (Participants) | 25
units on a scale | -3.84 (2.12)
Statistical Analysis 1: Comparison: Cingal; Test type: Other; p < 0.0001, ANOVA — P-Value was calculated

2. Secondary Outcome: American Orthopaedic Foot and Ankle Society (AOFAS) Score
Description: The change from baseline to 6 months in the American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Rating System, a standardized evaluation of the clinical status of the ankle-hindfoot. It incorporates both subjective and objective information in three parts to evaluate Pain, Function and Alignment. Patients report their pain (40 points), and function (50 points), and an evaluator assesses alignment (10 points). A total score is calculated by adding the three scores for a final range from 0 (worst clinical status) to 100 points (best clinical status).
  A positive increase in value for the change in AOFAS score indicates improvement. A larger positive value indicates a higher level of improvement, and a better outcome.
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cingal
Number analyzed (Participants) | 25
units on a scale | 15.88 (8.52)
Statistical Analysis 1: Comparison: Cingal; Test type: Other; p < 0.0001, ANOVA — P-Value was calculated

3. Secondary Outcome: Patient Global Assessment (PGA) Score
Description: The change from baseline to 6 months in ankle pain post-treatment as measured by the Patient Global Assessment (PGA) Score. PGA Score records participant responses to their assessment of how much their STUDY (treated) ankle is bothering them today . The PGA Score is a validated 11-point Likert scale ranged from 0 = No Pain to 10 = Worst Pain.
  A negative value for the change from baseline indicates improvement in PGA Score. A larger negative value indicates less pain, and a better clinical outcome.
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal
Number analyzed (Participants) | 25
score on a scale | -3.76 (2.01)
Statistical Analysis 1: Comparison: Cingal; Test type: Other; p < 0.0001, ANOVA — P-Value was calculated

4. Secondary Outcome: The Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index. A Calculated Percentage (%) of Participants Responding to Treatment.
Description: The post-treatment responder rate is determined through a calculation defined by the Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index. The OMERACT-OARSI Responder Index reports the percentage of subjects that met the criteria to be a good responder to treatment. The criteria for response are (1) improvement in pain or physical function >50% and an absolute change >20 mm; or (2) improvement of >20% with an absolute change >10 mm in at least of the following three categories: pain, physical function, and patient's global assessment.
  A higher percentage of subjects responding indicates a better outcome.
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Cingal
Number analyzed (Participants) | 25
Participants | 23

5. Secondary Outcome: Usage of Rescue Medication (Acetaminophen/Paracetamol). Number of Participants NOT Using Rescue Medication.
Description: The usage of Rescue Medication (RM) as based on the number of participants at 6 Months post treatment that were NOT using acetominophen/paracetamol RM for pain or discomfort.
  A larger percentage of participants that were NOT using RM may correlate to a better clinical outcome in terms of pain.
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Cingal
Number analyzed (Participants) | 25
Participants | 23

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of the Baseline Study Visit until Study Completion at 26 Weeks.
Description: The definitions of adverse events and serious adverse events is the same as used in the clinicaltrials.gov definitions.
  The incidence, timing, severity, and relationship to treatment of all Adverse Events (AE) were collected and coded using Medical Dictionary for Regulatory Activities (MedDRA).
Arm/Group | Cingal
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 4/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cingal (N=25)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 2 (2)

LIMITATIONS AND CAVEATS:
There were no limitations or caveats associated with the conduct of this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
INVESTIGATOR may publish the Data/Results with the consent of the SPONSOR if:

1. Publication is done after primary publication covering data from all participating sites, and provided the Data/Results do not contain any Confidential Information.
2. Eighteen (18) months has elapsed after entire completion of the Clinical Trial at all participating sites.

DOCUMENTS (2):
  • Study Protocol (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT04640974/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT04640974/SAP_001.pdf